CLINICAL TRIAL: NCT04706403
Title: If We Build It, Will They Come? A Pilot Study to Develop and Test Messages to Maximize Uptake of Coronavirus Vaccine When Available
Brief Title: Views on COVID-19 and Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Kimberly Fisher, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H00022244
Record Dates: First submitted 2021-01-05; First posted 2021-01-12 (Actual); Results first posted 2022-01-05 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Covid19
Keywords: Covid-19; Vaccination
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Message 1 (Experimental): Participants were randomized to receive version #1 of 5 different versions of a message from a physician regarding the COVID-19 vaccination. All messages included a statement that the vaccine is very safe and very effective. In Message 1, this statement was followed by a participatory-style recommendation ("What do you think?")
  Interventions: Behavioral: Communication from a physician about the COVID-19 Vaccine
- Message 2 (Experimental): Participants were randomized to receive version #2 of 5 different versions of a message from a physician regarding vaccination. All messages included a statement that the vaccine is very safe and very effective. In Message 2, this statement was followed by a comparison of the COVID-19 vaccine to the flu shot and an explicit recommendation ("I recommend that you get it").
  Interventions: Behavioral: Communication from a physician about the COVID-19 Vaccine
- Message 3 (Experimental): Participants were randomized to receive version #3 of 5 different versions of a message from a physician regarding vaccination. All messages included a statement that the vaccine is very safe and very effective. In Message 3, this statement was followed by a statement that millions of people have already received the COVID-19 vaccine and an explicit recommendation ("I recommend that you get it").
  Interventions: Behavioral: Communication from a physician about the COVID-19 Vaccine
- Message 4 (Experimental): Participants were randomized to receive version #4 of 5 different versions of a message from a physician regarding vaccination. All messages included a statement that the vaccine is very safe and very effective. In Message 4, this statement was followed by an acknowledgment of concerns and reassurance that the physician personally reviewed the safety data and an explicit recommendation ("I recommend that you get it").
  Interventions: Behavioral: Communication from a physician about the COVID-19 Vaccine
- Message 5 (Experimental): Participants were randomized to receive version #5 of 5 different versions of a message from a physician regarding vaccination. All messages included a statement that the vaccine is very safe and very effective. In Message 5, this statement was followed by an emphasis on protecting others an explicit recommendation ("I recommend that you get it").
  Interventions: Behavioral: Communication from a physician about the COVID-19 Vaccine

INTERVENTIONS:
Behavioral: Communication from a physician about the COVID-19 Vaccine — Participants who expressed hesitation about getting vaccinated against COVID-19 were randomized to receive one of five different versions of messages from a physician. The messages that participants in each group received varied slightly and systematically. Specific content and wording of these messages were developed to address and mitigate concerns of those at risk for not being vaccinated.

SUMMARY:
The goal of this study is to develop evidence-based messages that effectively mitigate concerns of people at risk for not being vaccinated against COVID-19, with the ultimate goal of maximizing vaccine uptake in vulnerable populations. The investigators will collect data on COVID-19 disease and vaccine knowledge, beliefs, and intent to be vaccinated from an existing online panel. Results from this data collection will be used to develop effective messages and communication strategies. The investigators will test alternate versions of messages intended to reduce vaccine hesitancy and promote vaccine uptake among vaccine-hesitant individuals. This project will ultimately result in a set of tested, evidence-derived messages about vaccination for COVID-19.

DETAILED DESCRIPTION:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has rapidly instigated a global pandemic. As of this writing, there are approximately 65 million documented cases of infection worldwide, and over 1.5 million deaths. In the United States (US), coronavirus disease 2019 (COVID-19) has disrupted the economy, overwhelmed healthcare system, led to widespread school cancellations, and caused more than 274,000 deaths since March 2020. A vaccine against COVID-19 is widely viewed as the key to controlling the pandemic and enabling a return to "normal" life. Vaccine development is proceeding at an unprecedented pace with 10 vaccines currently in phase 3 trials. Experts have projected that a safe and effective vaccine may be available by mid-2021. At the same time, a growing body of evidence indicates that a significant proportion of adults in the U.S. may not accept vaccination against COVID-19. Even more alarming, COVID-19 vaccine hesitancy (refusal or reluctance to accept a vaccine) appears to be increasing as the vaccine approval process becomes increasingly politicized. Just as efforts to develop vaccine production and delivery capacity have been undertaken in advance of having a proven effective vaccine, parallel efforts are needed to identify effective messages and communication strategies to overcome COVID-19 vaccine hesitancy.

The study team recently surveyed a nationally representative sample of approximately 1,000 adults in the United States and found that only 57% intended to be vaccinated when a coronavirus vaccine becomes available. This percentage was even lower among people who identified as Black or Hispanic (39% and 43% respectively), those with a high school education or less (46%), and those in the lowest income groups (49% of those reporting a household income of $30,000 or less, compared to 72% of those reporting a household income of $100,000 or more). The investigators asked those who indicated they would not or might not get vaccinated for their reasons and found that some individuals may be willing to be vaccinated if provided specific information about the vaccine such as side effects and effectiveness. Others expressed generalized skepticism, fear, and distrust of vaccines, with some even referring to anti-vaccine conspiracy theories. These findings are consistent with an extensive body of research documenting that people often do not behave rationally and highlight the urgent need to proactively develop and test interventions to maximize vaccination rates when a coronavirus vaccine becomes available. To address this need, in the present study, the investigators aim to create and test targeted messages to address the concerns of subgroups of people at risk for not being vaccinated, with the ultimate goal of maximizing vaccine uptake when a vaccine for COVID-19 becomes available. The investigators will accomplish this by working with an existing online panel of volunteers, which will allow efficient, focused data gathering. Results of the survey will provide a nuanced, current description of how vulnerable adults perceive the coronavirus and available vaccines, which will be used as the basis for developing messages and communication strategies. Participants will be randomized to receive one of five different versions of a message from a healthcare provider regarding vaccination. Specific wording and content of these messages will vary systematically in order to address concerns of those at risk for not being vaccinated. This project will ultimately result in a set of tested, evidence-derived messages about vaccination for COVID-19. The investigators will make these messages available, together with evidence of how these influence members of vulnerable populations' understanding of vaccination, and disease risk, as well as intent to be vaccinated. The messages will be freely available for use by organizations and providers seeking to improve communication about a coronavirus vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and over) who are members of an online panel (Prolific). Members of this panel joined the panel specifically to receive invitations to participate in research surveys and similar activities.
* Able to complete an online survey in English.

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Fisher, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Meyers Health Care Institute, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher KA, Bloomstone SJ, Walder J, Crawford S, Fouayzi H, Mazor KM. Attitudes Toward a Potential SARS-CoV-2 Vaccine : A Survey of U.S. Adults. Ann Intern Med. 2020 Dec 15;173(12):964-973. doi: 10.7326/M20-3569. Epub 2020 Sep 4. PMID 32886525
- [Background] Brewer NT, Chapman GB, Rothman AJ, Leask J, Kempe A. Increasing Vaccination: Putting Psychological Science Into Action. Psychol Sci Public Interest. 2017 Dec;18(3):149-207. doi: 10.1177/1529100618760521. PMID 29611455
- [Background] Godinho CA, Yardley L, Marcu A, Mowbray F, Beard E, Michie S. Increasing the intent to receive a pandemic influenza vaccination: Testing the impact of theory-based messages. Prev Med. 2016 Aug;89:104-111. doi: 10.1016/j.ypmed.2016.05.025. Epub 2016 May 25. PMID 27235605
- [Background] Mowbray F, Marcu A, Godinho CA, Michie S, Yardley L. Communicating to increase public uptake of pandemic flu vaccination in the UK: Which messages work? Vaccine. 2016 Jun 14;34(28):3268-74. doi: 10.1016/j.vaccine.2016.05.006. Epub 2016 May 8. PMID 27166824
- [Background] Nowak GJ, Sheedy K, Bursey K, Smith TM, Basket M. Promoting influenza vaccination: insights from a qualitative meta-analysis of 14 years of influenza-related communications research by U.S. Centers for Disease Control and Prevention (CDC). Vaccine. 2015 Jun 4;33(24):2741-56. doi: 10.1016/j.vaccine.2015.04.064. Epub 2015 Apr 28. PMID 25936726
- [Background] Redelings MD, Piron J, Smith LV, Chan A, Heinzerling J, Sanchez KM, Bedair D, Ponce M, Kuo T. Knowledge, attitudes, and beliefs about seasonal influenza and H1N1 vaccinations in a low-income, public health clinic population. Vaccine. 2012 Jan 5;30(2):454-8. doi: 10.1016/j.vaccine.2011.10.050. Epub 2011 Oct 30. PMID 22044740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited on Prolific.co from 01/12/21-02/01/21. Eligible panel members were >= 18, English speaking, and U.S residents. Panel members were restricted to include White, Black, or Hispanic; Blacks and Hispanics were oversampled. Participants who responded "no" or "not sure" to "If you could get vaccinated for COVID-19 today, would you?" were classified as vaccine hesitant and randomized to receive 1 of 5 physician messages, after which their intent was reassessed.
Period: Overall Study
Arm/Group | Message 1 | Message 2 | Message 3 | Message 4 | Message 5
Started | 172 | 121 | 165 | 146 | 152
Completed | 172 | 121 | 164 | 145 | 150
Not Completed | 0 | 0 | 1 | 1 | 2
Not completed — Participants did not provide respond to the question re-assessing vaccination intent | 0 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Message 4: Participants were randomized to receive version #4 of 5 different versions of a message from a physician regarding vaccination. All messages included a statement that the vaccine is very safe and very effective. In Message 4, this statement was followed by an acknowledgement of concerns and reassurance that the physician personally reviewed the safety data and an explicit recommendation ("I recommend that you get it").
- Total: Total of all reporting groups
Arm/Group | Message 1 | Message 2 | Message 3 | Message 4 | Message 5 | Total
Number analyzed (Participants) | 172 | 121 | 164 | 145 | 150 | 752
Age, Customized [Count of Participants; unit: Participants]
  Age: Less than 24 years | 43 | 31 | 37 | 38 | 41 | 190
  Age: 25 - 34 years | 40 | 32 | 42 | 28 | 42 | 184
  Age: 35 - 44 years | 50 | 27 | 31 | 50 | 33 | 191
  Age: 45 - 54 years | 22 | 21 | 27 | 17 | 20 | 107
  Age: 55 - 64 years | 13 | 4 | 20 | 10 | 11 | 58
  Age: 65 years or older | 3 | 5 | 3 | 2 | 2 | 15
  Age: Missing | 1 | 1 | 4 | 0 | 1 | 7
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 62 | 41 | 71 | 52 | 65 | 291
  Gender: Female | 108 | 78 | 88 | 93 | 82 | 449
  Gender: Other | 0 | 2 | 4 | 0 | 0 | 6
  Gender: Prefer not to say | 1 | 0 | 0 | 0 | 0 | 1
  Gender: Missing | 1 | 0 | 1 | 0 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 35 | 31 | 41 | 33 | 37 | 177
  Black/African American | 79 | 52 | 66 | 64 | 65 | 326
  White | 58 | 37 | 57 | 48 | 48 | 248
  Missing | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 172 | 121 | 164 | 145 | 150 | 752
Initial Vaccination Intent [Count of Participants; unit: Participants]
  Initially "No" | 103 | 66 | 83 | 78 | 81 | 411
  Initially "Not Sure" | 69 | 55 | 81 | 67 | 69 | 341
Education [Count of Participants; unit: Participants]
  High School or Less | 44 | 40 | 53 | 38 | 49 | 224
  Some college | 86 | 56 | 85 | 70 | 68 | 365
  4-year college or more | 42 | 25 | 25 | 36 | 32 | 160
  Missing | 0 | 0 | 1 | 1 | 1 | 3
Employment [Count of Participants; unit: Participants]
  Employed | 88 | 64 | 83 | 83 | 76 | 394
  Unemployed | 30 | 20 | 29 | 20 | 30 | 129
  Student | 25 | 15 | 15 | 19 | 18 | 92
  Homemaker | 16 | 12 | 9 | 14 | 13 | 64
  Disabled | 6 | 3 | 10 | 4 | 5 | 28
  Retired | 3 | 3 | 7 | 4 | 4 | 21
  Other | 4 | 3 | 10 | 1 | 4 | 22
  Missing | 0 | 1 | 1 | 0 | 0 | 2
Household Income [Count of Participants; unit: Participants]
  Less than $30,000 | 47 | 43 | 55 | 40 | 57 | 242
  $30,000 - $60,000 | 53 | 41 | 57 | 51 | 53 | 255
  $60,000 - $100,000 | 44 | 27 | 35 | 26 | 27 | 159
  More than $100,000 | 21 | 7 | 11 | 19 | 9 | 67
  Prefer not to answer | 6 | 2 | 5 | 9 | 3 | 25
  Missing | 1 | 1 | 1 | 0 | 1 | 4
Geographic region [Count of Participants; unit: Participants]
  South | 90 | 66 | 80 | 75 | 80 | 391
  Midwest | 28 | 17 | 34 | 31 | 21 | 131
  West | 28 | 21 | 23 | 15 | 33 | 120
  Northeast | 26 | 17 | 27 | 24 | 16 | 110
History of flu shot [Count of Participants; unit: Participants]
  Ever, in the last 5 years | 73 | 40 | 70 | 78 | 71 | 332
  Not sure or no | 99 | 81 | 93 | 67 | 79 | 419
  Missing | 0 | 0 | 1 | 0 | 0 | 1
Self-rated overall health [Count of Participants; unit: Participants]
  Excellent | 22 | 12 | 13 | 9 | 13 | 69
  Very good | 44 | 34 | 48 | 40 | 39 | 205
  Good | 69 | 51 | 66 | 58 | 65 | 309
  Fair | 27 | 19 | 34 | 33 | 24 | 137
  Poor | 9 | 5 | 3 | 5 | 8 | 30
  Missing | 1 | 0 | 0 | 0 | 1 | 2
Self-rated overall mental health [Count of Participants; unit: Participants]
  Excellent | 22 | 17 | 22 | 12 | 18 | 91
  Very good | 43 | 31 | 37 | 33 | 30 | 174
  Good | 42 | 38 | 48 | 47 | 50 | 225
  Fair | 51 | 20 | 39 | 35 | 40 | 185
  Poor | 14 | 15 | 18 | 17 | 12 | 76
  Missing | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Became Less Hesitant About the COVID-19 Vaccine After Receiving a Physician Message
Description: All participants were asked about their intent to be vaccinated against COVID-19 prior to exposure to one of the five physician messages (Response options: Yes, No, Not sure). After participants were randomly assigned to receive one of the five physician messages, reduction in COVID-19 vaccine hesitancy was assessed with the question: "Would you get vaccinated at this visit". Response options included yes, no, not sure. For participants whose initial vaccination intent was "not sure", a response of "yes" on re-assessment was defined as less hesitant. Response of "not sure" or "yes" were defined as less hesitant for participants whose initial vaccination intent was "no".
Time Frame: Through survey completion, an average of 12 minutes
Population: Four participants were excluded from the analyses because they did not respond to the question re-assessing vaccination intent following exposure to a physician recommendation.
Measure: Count of Participants; unit: Participants
Arm/Group | Message 1 | Message 2 | Message 3 | Message 4 | Message 5
Number analyzed (Participants) | 172 | 121 | 164 | 145 | 150
Participants | 23 | 26 | 43 | 35 | 40

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- Message 4: Participants were be randomized to receive version #4 of 5 different versions of a message from a physician regarding vaccination. All messages included a statement that the vaccine is very safe and very effective. In Message 4, this statement was followed by an acknowledgment of concerns and reassurance that the physician personally reviewed the safety data and an explicit recommendation ("I recommend that you get it").
Arm/Group | Message 1 | Message 2 | Message 3 | Message 4 | Message 5
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Limitations include: (1) Inability to assess whether the impact of physician messages in practice would parallel the impact in the hypothetical scenarios used in this study; (2) The use of an online research platform (prolific.co) may limit generalizability of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT04706403/Prot_SAP_000.pdf